CLINICAL TRIAL: NCT00002656
Title: PHASE II CLINICAL EVALUATION OF PYRAZOLOACRIDINE IN PATIENTS WITH ADVANCED NON-SMALL CELL LUNG CARCINOMA
Brief Title: Pyrazoloacridine in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000064199; P30CA022453 (NIH); WSU-C-1087-93; NCI-T94-0001H
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — NSC 366140

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pyrazoloacridine (Experimental): Pyrazoloacridine 750 mg/m2 by 3 hour infusion, every 21 day s in the absence of progressive disease or prohibitive toxicity.
  Interventions: Drug: pyrazoloacridine

INTERVENTIONS:
Drug: pyrazoloacridine — Pyrazoloacridine 750 mg/m2 by 3 hour infusion, every 21 day s in the absence of progressive disease or prohibitive toxicity.
  Depending on the prior cycle toxicity the dose should be escalated, maintained or reduced, utilizing levels: -1, 0 (initial dose level), 1 - Level +1 (820mg/m2); Level 0 (750mg/m2); Level -1 (600mg/m2)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy with pyrazoloacridine in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the antitumor activity of pyrazoloacridine (PZA) administered by 3-hour infusion to patients with advanced non small cell lung cancer (NSCLC). II. Determine the qualitative and quantitative toxicities of PZA administered on this schedule. III. Determine the response and survival durations of NSCLC patients treated with PZA.

OUTLINE: Single-Agent Chemotherapy. Pyrazoloacridine, PZA, NSC-366140.

PROJECTED ACCRUAL: If 2 or 3 responses are observed in the first 18 evaluable patients, 12 additional patients will be entered. Accrual is expected to take 5-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed non small cell lung cancer ineligible for higher priority protocols Sputum cytology acceptable Stage IIIB/IV Must have measurable or evaluable disease Lesion outside prior radiotherapy fields Cytology-positive pleural effusion and ascites are neither measurable nor evaluable No brain metastases on CT

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count greater than 2,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL Renal: Creatinine less than 1.5 mg/dL Other: No pregnant or nursing women Negative pregnancy test required of fertile women Effective contraception required of fertile patients Blood/body fluid analyses within 7 days prior to registration Imaging/exams for tumor measurement within 28 days prior to registration

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: One prior adjuvant or neoadjuvant chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since radiotherapy and recovered AND Progressive disease outside of radiation port Surgery: Recovered from any prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1995-10; Primary Completion 2001-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Evaluate toxicity of pyrazoloacridine. | Weekly prior to each treatment cycle.

SECONDARY OUTCOMES:
Evaluate the response frequency of pyrazoloacridine. | After 2 treatment cycles then every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette J. Wozniak, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States